CLINICAL TRIAL: NCT06198803
Title: The Effect of Carnitine Supplementation on Cardiac Function and Lipid Profile in Patients With Drug Resistant Epilepsy on Ketogenic Diet
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: carnitine effect on cardiac
Record Dates: First submitted 2023-11-02; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-10

CONDITIONS: l Carnitine With Ketogenic Diet
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: All aged from 1 month till 16 years old with DRE on KD.
Who Masked: Participant
Masking Description: Patients who are already on KD and carnitine supplements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- l carnitine group (Experimental): All aged from 1 month till 16 years old with DRE on KD.
  Interventions: Drug: L Carnitine
- non l carnitine gruop (No Intervention): patient with drug resistant epilepsy on ketogenic diet

INTERVENTIONS:
Drug: L Carnitine — The study population will be randomly divided into 2 groups, 1 group will receive Carnitine supplementation in a dose of 100mg/kg/day
  Arms: l carnitine group

SUMMARY:
Primary aim: Demonstrating the effect of carnitine supplementation on lipid profile and cardiovascular functions in patients with DRE on KD.

Secondary aim: To highlight the effect of carnitine supplementation on efficacy of KD in seizure control.

DETAILED DESCRIPTION:
The KD, a strict diet high in fat and low in carbohydrates, increases the ketone body concentrations that could lead to an enhancement of inhibitory neurotransmission and thereby possibly reducing the seizure frequency (Seo et al., 2007).

Carnitine plays a major role in the degradation of fatty acids. As a trimethylated amino acid, it facilitates translocation of fatty acids into the mitochondrion and is therefore an essential cofactor in fatty acid oxidation and ketogenesis (Longo et al., 2016).

Carnitine transports dietary fat to the mitochondria to be oxidized into ketones, which are used for energy when sufficient carbohydrate is not available (Coppola et al., 2006; Mcnally & Hartman, 2012).

Levocarnitine can improve cardiac function effectively through improving albumin, high sensitivity CRP, Brain natriuretic protein, troponin, and left ventricular end diastolic dimension (Zhao et al., 2020).

Due to the high fat intake, children following KD may have an increased demand for carnitine and therefore, may be at an increased risk for carnitine deficiency (Neal EG et al.,2008).

Although total carnitine decrease over the first few months of KD treatment, and in some patients, dip into the deficiency range, it then normalizes with no evidence of a continued decline (Berry-Kravis et al., 2001; Coppola et al., 2006).

Few studies was performed to evaluate carnitine effect in epileptic children and adolescents treated with old and new antiepileptic drugs with or without ketogenic diet Coppola et al., 2006).

The KD is mostly associated with Gastrointestinal (GI) disturbances, such as nausea, vomiting, diarrhea, and constipation, also were frequently noted, sometimes associated with gastritis and fat intolerance (Armeno et al., 2018).

ELIGIBILITY:
Inclusion Criteria:

- All aged from 1 month till 16 years old with DRE on KD.

Exclusion Criteria:

* Patients who are already on KD and carnitine supplements.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The Effect of Carnitine Supplementation on systolic and diastolic functions in Patients With Drug Resistant Epilepsy on Ketogenic Diet | baseline
  Demonstrate The effect of carnitine supplementation on Ejection Fraction to assess systolic and E/A ratio to assess diastolic functions in patients with drug resistant epilepsy on Ketogenic Diet
The Effect of Carnitine supplementation on serum triglycerides, cholesterol, LDL and HDL in lipid profile in Patients With Drug Resistant Epilepsy on Ketogenic Diet | baseline
  the effect of carnitine supplementation on serum triglycerides in milligrams per deciliter, cholesterol in milligrams per deciliter, LDLin milligrams per deciliter and HDL in milligrams per deciliter in lipid profile in patients with drug resistant epilepsy on ketogenic diet
The Effect of Carnitine supplementation on Convulsions in Patients With Drug Resistant Epilepsy on Ketogenic Diet | baseline
  the effect of carnitine supplementation on chalfont seizure severity scale to assess convulsions in patients with drug resistant epilepsy on ketogenic diet

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo, Cairo, Egypt